CLINICAL TRIAL: NCT04973917
Title: A Prospective Comparison of the Efficacy and Safety of Intellectual Mode of Ventilation (Intellivent-ASV) With Conventional Modes in Cardiac Surgery Patients With Body Mass Index >35
Brief Title: A Comparison of Intellivent-ASV Mode With Conventional Modes in Patients With BMI >35
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13120001
Record Dates: First submitted 2021-06-24; First posted 2021-07-22 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Ventilation Therapy; Complications
Keywords: postoperative care; closed-loop modes; safety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional ventilation mode (Experimental): respiratory support after cardiac surgery. Vt < 6 ml/kg PBW, driving pressure < 13 cmH2O
  Interventions: Procedure: respiratory support
- intelectual mode - Intelivent ASV (Experimental): closed loop mode of mechanical ventilation Vt < 6 ml/kg PBW, driving pressure < 13 cmH2O
  Interventions: Procedure: respiratory support

INTERVENTIONS:
Procedure: respiratory support — respirators for invasive mechanical ventilation

SUMMARY:
compare effects of intellectual mode (in our case it will be Intellivent - ASV -) with conventional ventilation modes after uncomplicated cardiac surgery in patients with body mass index >35

DETAILED DESCRIPTION:
The study includes the comparison of two methods of invasive respiratory support ventilation( conventional ventilation modes and automatic IntelliventASV mode (a fully automated, or closed-loop, ventilation mode that consists of pressure-controlled ventilation or pressure support ventilation depending on a patient's respiratory activity. In fully automated ventilation mode, tidal volume, pressure levels (including PEEP), minute ventilation, and the oxygen fraction in inspired air are controlled solely by the ventilator) after uncomplicated cardiac surgery). It assumes 30 randomized patients:15 patients in two study groups male and female aged 30 to 70 years of age inclusive, with BMI > 35 kg/m2. The study will be randomized, single-center, prospective.

ELIGIBILITY:
Inclusion Criteria:

* • Age from 30 years to 70 years inclusive

  * elective cardiac surgery which included bypass, valve and ascending aortic surgery,
  * a body mass index of > 35 kg/m2,
  * postoperative treatment with mechanical ventilation,
  * informed consent

Exclusion Criteria:

* • GFI <30 ml/min before surgery, serum aspartate and alanine transaminase concentration greater than 80 U/l before surgery, left ventricular ejection fraction less than 30% before surgery.

Postoperative exclusion criteria:

* chest tube drainage greater than 3 ml/kg/h,
* reoperation,
* myocardial infarction,
* need for high-dose inotropes or vasopressors or intraaortic balloon pump,
* presence of a bronchopleural fistula and refractory hypoxemia with an arterial oxygen tension to fractional inspired oxygen concentration ratio less than 150 mmHg,
* perioperative anaphylactic reaction,
* seizures,
* stroke,
* agitation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with tidal volume in optimal, suboptimal, unoptimal zone | During the first 8 hours, since admission on the ICU with the start of the respiratory support
  Number of Participants during mechanical ventilation with Tidal volume in optimal zone < 6 ml/kg/Predicted Body Weight ; Tidal volume in suboptimal zone 6-8 ml/kg/Predicted Body Weight Tidal volume in unoptimal zone >8 ml/kg/Predicted Body Weight

SECONDARY OUTCOMES:
the physician's workload | 24 hours
  accounting number of manual ventilator settings changes made before extubation of trachea

CONTACTS AND LOCATIONS:
Overall Officials: Alexandr Eremenko, Professor, Principal Investigator — Russian research center of surgery named after B. V. Petrovsky
Locations (1):
- Russian research center of surgery named after academician B. V. Petrovsky, Moscow, Г. Москва, Russia

IPD SHARING:
Plan to Share IPD: No